CLINICAL TRIAL: NCT04992455
Title: The Predictive Value of G8, VES-13 and CARG Scores in Treatment-related Toxicity in Geriatric Cancer Patients
Brief Title: G8, VES-13 and CARG Scores in Predicting Chemotherapy Toxicity in Geriatric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Asoc. Prof. Erdoğan Selçuk Şeber, assoc prof, Namik Kemal University
Other Study IDs: CHEMOTOXTOOL
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Predicting Chemotherapy Related Toxicity in Elderly Patients
Keywords: g8; ves-13; CARG; chemotherapy-related toxicity; Toxicity tool

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Older Patients Receiving Chemotherapy — No Intervention

SUMMARY:
All participants' medical information will be collected for use as a baseline, including tumor-specific variables, nutritional status, functional status, psychological status, cognitive function, social support, and comorbidities. The suitability of G8, VES-13 and CARG chemotherapy risk assessment tools for elderly cancer patients was investigated.

DETAILED DESCRIPTION:
All participants' medical information will be collected for use as a baseline, including tumor-specific variables, nutritional status, functional status, psychological status, cognitive function, social support, and comorbidities. G8, VES-13 and CARG toxicity scores of all participating patients will be determined by two independent investigators before starting chemotherapy. The suitability of these practical chemotherapy risk assessment tools for cancer patients for elderly cancer patients was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years
* Localized or metastatic solid carcinoma diagnosed by histology (any type, any stage)
* Starting a new-line (first-line, second-line or third-line) chemotherapy

Exclusion Criteria:

* Concurrent radiotherapy;
* Simultaneous immunotherapy
* Impaired language
* Cognitive function leading to inability to complete assessments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older Patients Receiving Chemotherapy
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
G8 (Geriatric 8) screening tool measurement | 15-30 minutes
CARG (Cancer and Aging Research Group) chemotherapy toxicity score measurement | 30-60 minutes
VES-13 (Vulnerable Elders Survey-13) measurement | 30-60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Erdoğan S Şeber, Assoc. Prof., Study Chair — Namik Kemal University; Eyyüp Çavdar, MD, Study Director — Namik Kemal University
Locations (1):
- Tekirdağ Namık Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided